CLINICAL TRIAL: NCT05351307
Title: Retinal Vascular Changes in Primary Open Angle Glaucoma Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marwa Hamza Ali, Principal investigator, Sohag University
Other Study IDs: Soh-Med-22-03-03
Record Dates: First submitted 2022-04-24; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POAG patients: OCT angiography will be performed
- Normal participants: OCT angiography will be performed

SUMMARY:
the study aims to detect ischemic changes in macula using OCT angiography in primary open angle glaucoma patients correlating with glaucoma staging system II by visual field.

DETAILED DESCRIPTION:
Our study will be designed as " prospective non-randomized case - control study" The study will include 100 eyes of 100 participants 50 eyes of normal subjects , non-glaucomatous subjects 50 eyes of 50 patients with POAG To detect ischemic changes in macula using OCT angiography correlating with glaucoma staging system II by visual field.

ELIGIBILITY:
Inclusion Criteria:

* (> 18 years old)

Exclusion Criteria:

* patients with cataract
* retinal disorders including: AMD , Macular degeneration , retinal detachment , retinitis pigmentosa , etc .
* corneal opacites
* any ocular surgeries
* patients with systemic disease.
* patient refusal

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: > 18 years primary open angle glaucoma patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
ischemic changes in macula | Through one year
  Using OCT angiography to detect ischemic changes in macula

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Iqbal Hafez, Assist prof, Study Director — Supervisor; Hany Mahmoud Abdel Hamid, Lecturer, Study Director — Supervisor
Locations (1):
- Sohag University hospitals, Sohag, Egypt